CLINICAL TRIAL: NCT04172584
Title: Awareness & Use of Emergency Contraception Among Women Attending Kidwany MCH Center , Assiut City
Brief Title: Awareness & Use of Emergency Contraception
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marian Agaiby Ashem, Doctor, Assiut University
Other Study IDs: Emergency contraception.
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Emergency Contraception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: correct use of the contraceptions — know the emergency contraception and how to use

SUMMARY:
General objective:

To decrease the percentage of unwanted and/or unplanned pregnancies and their consequences on women's reproductive health.

Specific objectives:

1. To assess awareness of the study participants about emergency contraception.
2. Determine the percentage of ever use among the participants.
3. To identify factors that affect the awareness and use of emergency contraception among the study participants

ELIGIBILITY:
Inclusion Criteria:

* Married women in reproductive age (15 - 49 years)

Exclusion Criteria:

* Infertile and postmenopausal women.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Married women in reproductive age (15 - 49 years) clients who are attending Kidwany MCH centre, Assiut city.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent of awareness and use of emergency contraception | baseline
  when to use emergency contraception to prevent the unwanted pregnancy

REFERENCES:
- [Background] Mohammed S, Abdulai AM, Iddrisu OA. Pre-service knowledge, perception, and use of emergency contraception among future healthcare providers in northern Ghana. Contracept Reprod Med. 2019 Jan 24;4:1. doi: 10.1186/s40834-018-0082-9. eCollection 2019. PMID 30693098
- [Result] Mittal S. Emergency contraception: which is the best? Minerva Ginecol. 2016 Dec;68(6):687-99. Epub 2016 Apr 15. PMID 27082029
- [Result] Association of Women's Health, Obstetric and Neonatal Nurses. Emergency Contraception. J Obstet Gynecol Neonatal Nurs. 2017 Nov-Dec;46(6):886-888. doi: 10.1016/j.jogn.2017.09.004. No abstract available. PMID 29128088